CLINICAL TRIAL: NCT02210416
Title: Costs of Complications in Inguinal Hernia Repair
Status: Completed | Type: Observational
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Kouhia, MD, North Karelia Central Hospital
Other Study IDs: NKCH-Surg-011
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Inguinal Hernia; Complication
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LAP repair: patients receiving laparoscopic inguinal hernia repair
  Interventions: Procedure: inguinal hernia surgery
- open repair: patients receiving open flat mesh repair of inguinal hernia
  Interventions: Procedure: inguinal hernia surgery

INTERVENTIONS:
Procedure: inguinal hernia surgery

SUMMARY:
Laparoscopic inguinal hernia repair is becoming increasingly popular mainly because of short-term advantages compared to open hernioplasties with mesh. In the prevailing economic climate, the total costs of treatment is a subject of intense research. This study is designed to evaluate the results of open and laparoscopic inguinal hernia repairs, with a special emphasis in costs of treatment, complications and convalescence.

ELIGIBILITY:
Inclusion Criteria:

* patients treated surgically for inguinal hernia between 2002-2011

Exclusion Criteria:

* none

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing laparoscopic inguinal hernia repair (TAPP or TEP) during 2002-2011 A sample of 528 patients undergoing open flat mesh repair in 2002-2011.
Sampling Method: Non-Probability Sample
Enrollment: 968 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
cost of complication | 3 years
  any complication associated with hernia surgery within 3 years, and its total costs
cost of primary treatment | 2 months
  the in-hospital costs of inguinal hernia repair surgery and the costs of convalescence following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- North Karelia Central Hospital, Joensuu, Finland